CLINICAL TRIAL: NCT07401030
Title: The Effectiveness of a Psychological Resilience Training Program for Children Aged 10-12: An Evaluation in Terms of Psychological Resilience, Social Adjustment, Close Relationships, and Media Use
Brief Title: Effectiveness of a Psychological Resilience Training Program for Children Aged 10-12
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yusuf AKTEPE (Other)
Responsible Party: Sponsor-Investigator, Yusuf AKTEPE, Principal Investigator and MSc Researcher, Agri Ibrahim Cecen University
Organization: Agri Ibrahim Cecen University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: AICU-SBF-YA-01
Record Dates: First submitted 2026-02-02; First posted 2026-02-10 (Actual); Last update posted 2026-02-10 (Actual); Status verified 2026-02

CONDITIONS: Psychological Resilience; Social Adjustment; Interpersonal Relationships; Media Use
Keywords: Psychological Resilience; Resilience Training Program; Children Aged 10-12; Social Adjustment; Interpersonal Relationships; Parent-Child Relationship; Problematic Media Use; School-Based Intervention; Randomized Controlled Trial
MeSH Terms: conditions — Social Adjustment

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to either an intervention group or a control group and will remain in their assigned group for the entire duration of the study. The intervention and control groups will proceed in parallel and will not cross over or switch interventions at any point.
Who Masked: Outcomes Assessor
Masking Description: Outcome assessors and data analysts will be blinded to group allocation. Participants are not blinded due to the nature of the intervention.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Psychological resilience training program (Experimental): Participants in this arm will receive a structured psychological resilience training program designed for children aged 10-12 years. The program will be delivered in a group format and will consist of 10 sessions over a five-week period. The sessions will focus on emotion recognition and regulation, self-awareness, self-efficacy, coping with stress, problem-solving skills, social skills, social support, and media use awareness.
  Interventions: Behavioral: Psychological Resilience Training Program
- No-intervention control (No Intervention): Participants in this arm will not receive any psychological or educational intervention during the study period. They will continue with their usual school activities and will complete the same assessments as the intervention group at the scheduled time points.

INTERVENTIONS:
Behavioral: Psychological Resilience Training Program — This is a structured, school-based psychological resilience training program designed for children aged 10-12 years. The program consists of 10 group sessions delivered over a five-week period (two sessions per week). Session content includes emotion recognition and regulation, self-awareness and identification of personal strengths, self-efficacy, coping with stressful situations, problem-solving skills, cognitive flexibility, social skills development, communication skills, social support utilization, and media use awareness and self-control.
  Arms: Psychological resilience training program

SUMMARY:
This clinical study aims to learn whether a psychological resilience training program is helpful for children aged 10 to 12 years. The program is designed to help children cope better with stress, get along better with others, and use digital media in a healthier way.

The main questions this study seeks to answer are:

Does the training increase children's psychological resilience?

Does it improve children's social adjustment and close relationships with family and friends?

Does it help reduce problematic media use?

Children who take part in the study are randomly assigned to one of two groups. One group takes part in a psychological resilience training program, and the other group does not receive any training during the study period. Children and their parents complete questionnaires before the program and again after the program is completed.

DETAILED DESCRIPTION:
This study is planned as a randomized controlled interventional trial to evaluate the effects of a structured psychological resilience training program on multiple psychosocial outcomes in children aged 10-12 years. The study will be conducted in a school setting in Agri, Turkey.

A total of 50 eligible children who meet the inclusion criteria will be enrolled in the study. After completion of baseline assessments, participants will be randomly assigned to an intervention group (n = 25) or a control group (n = 25) using a simple randomization method. Group allocation will be coded to reduce potential bias during data analysis. Participants and their parents will not be informed about group assignment, and statistical analyses will be performed by an independent analyst who will be blinded to group codes.

The intervention group will receive a school-based psychological resilience training program developed for children and adolescents. The program will be delivered in a group format and will consist of 10 sessions implemented over a five-week period, with two sessions per week. The session content will include emotional awareness and regulation, self-awareness and identification of personal strengths, self-efficacy, coping with stressful situations, problem-solving skills, cognitive flexibility, social skills development, communication skills, utilization of social support resources, and media use awareness and self-control. The control group will not receive any intervention during the study period and will participate only in assessment procedures.

Data will be collected at two time points: at baseline (prior to randomization) and at follow-up after completion of the intervention period. Child-reported and parent-reported standardized measures will be used to assess psychological resilience, social adjustment, problematic media use, and parent-child relationship characteristics. The study will be conducted in accordance with ethical principles and will be approved by a university ethics committee prior to participant enrolment.

ELIGIBILITY:
Inclusion Criteria:

* Children aged 10 to 12 years
* Enrollment in a primary or middle school
* Ability to understand and participate in group-based educational activities
* Willingness of the child to participate in the study
* Written informed consent provided by a parent or legal guardian
* No prior participation in a psychological resilience or emotional regulation training program

Exclusion Criteria:

* Presence of a diagnosed severe psychiatric disorder (e.g., psychotic disorders or severe behavioral disorders)
* Cognitive impairment that would prevent understanding the training content or completing assessments
* Participation in another psychological or behavioral intervention during the study period
* Absence from a substantial portion of the intervention sessions
* Withdrawal of consent by the child or parent/legal guardian at any stage of the study

Ages: 10 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 50 (Estimated)
Dates: Start 2026-02-02 (Estimated); Primary Completion 2026-03-20 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
PSYCHOLOGICAL RESILIENCE | Time Frame: Baseline (before the intervention) and follow-up (one month after completion of the training program)
  Psychological resilience will be measured using the Children and Youth Resilience Measure-12 (CYRM-12). This scale assesses children's ability to cope with stress and challenging life situations. Total scores range from 12 to 60, with higher scores indicating greater psychological resilience.

SECONDARY OUTCOMES:
SOCIAL ADJUSTMENT | Time Frame: Baseline (before the intervention) and follow-up (one month after completion of the training program)
  Social adjustment will be measured using the Social Adjustment Scale (SUÖ). This scale assesses children's ability to adapt to social rules, interact effectively with peers, and function appropriately in social settings. Total scores range from 55 to 275, with higher scores indicating better social adjustment.
PROBLEMATIC MEDIA USE | Time Frame: Baseline (before the intervention) and follow-up (one month after completion of the training program)
  Problematic media use will be assessed using the Problematic Media Use Scale (PMKÖ), a parent-reported measure that evaluates children's difficulties in controlling and regulating digital media and screen use. Scores are calculated on a Likert-type scale ranging from 1 to 5, with higher scores indicating more problematic media use.
PARENT-CHILD RELATIONSHIP | Time Frame: Baseline (before the intervention) and follow-up (one month after completion of the training program)
  Parent-child relationship will be assessed using the Parent-Child Relationship Scale (EÇİÖ), a parent-reported instrument consisting of 15 items that assess both positive and negative dimensions of the parent-child relationship. Items are rated on a 5-point Likert scale ranging from 1 (not at all) to 5 (extremely). Higher scores on the positive subscale indicate more positive relationship characteristics, whereas higher scores on the negative subscale indicate more negative relationship characteristics.

CONTACTS AND LOCATIONS:
Overall Officials: Yusuf AKTEPE, MSc / RN / Graduate Student, Principal Investigator — Agri Ibrahim Cecen University
Locations (1):
- Alpaslan Middle School, Ağrı, Ağrı, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared. The study involves minors, and data include sensitive personal and psychological information collected under ethical approval and informed consent that do not permit public data sharing.

REFERENCES:
- [Background] Masten AS. Resilience in children threatened by extreme adversity: Frameworks for research, practice, and translational synergy. Development and Psychopathology. 2011;23(2):493-506.